CLINICAL TRIAL: NCT03183921
Title: Epidemiological, Microbiological and Clinical Profile of Ice Patients With Nosocomial Lower Respiratory Tract Infections
Brief Title: Study on ICU Patients With Nosocomial Lower Respiratory Tract Infections
Acronym: ENIRRIs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: ENIRRIs 01
Record Dates: First submitted 2017-04-20; First posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: All ICU patients with nosocomial lower respiratory tract infection
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Interventions

SUMMARY:
This is a multicentre, multinational, prospective observational investigation on ICU critically ill patients affected by nosocomial pneumonia, defined as: Out of ICU Hospital-acquired Pneumonia (HAP), Non-ventilator ICU-acquired Pneumonia (NV ICUAP), Ventilator associated pneumonia (VAP) Ventilator associated tracheobronchitis (VAT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of nosocomial pneumonia
* ICU and HDU admission (patient may be admitted to the ICU with NP or may develop pneumonia during ICU stay)
* Informed consent (if required)

Exclusion Criteria:

* Community Acquired Infection
* Absence of Microbiological Findings

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ICU patients with a documented Nosocomial Lower Respiratory Tract Infection will be eligible for this epidemiological, clinical and microbiological investigation
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients dying among the different pneumonia categories | 28 days

SECONDARY OUTCOMES:
Number of patients with different epidemiological patterns | 28 days
Number of patients with specific microbiological profiles | 28 days
Number of patients with specific clinical characteristics | 28 days
Number of patients with different therapeutically interventions | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- St James's University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Martin-Loeches I, Reyes LF, Nseir S, Ranzani O, Povoa P, Diaz E, Schultz MJ, Rodriguez AH, Serrano-Mayorga CC, De Pascale G, Navalesi P, Panigada M, Coelho LM, Skoczynski S, Esperatti M, Cortegiani A, Aliberti S, Caricato A, Salzer HJF, Ceccato A, Civljak R, Soave PM, Luyt CE, Ekren PK, Rios F, Masclans JR, Marin J, Iglesias-Moles S, Nava S, Chiumello D, Bos LD, Artigas A, Froes F, Grimaldi D, Taccone FS, Antonelli M, Torres A; European Network for ICU-Related Respiratory Infections (ENIRRIs) European Respiratory Society-Clinical Research Collaboration Investigators. European Network for ICU-Related Respiratory Infections (ENIRRIs): a multinational, prospective, cohort study of nosocomial LRTI. Intensive Care Med. 2023 Oct;49(10):1212-1222. doi: 10.1007/s00134-023-07210-9. Epub 2023 Oct 9. PMID 37812242